CLINICAL TRIAL: NCT04369079
Title: Myofascial Versus Conventional Physiotherapy in Post-mastectomy Patients: a Randomized Controlled Trial
Brief Title: Myofascial Versus Conventional Physiotherapy
Acronym: MYONAMASTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Greater Poland Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MYONAMASTE
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-04

CONDITIONS: Sports; Therapy
Keywords: physiotherapy; Myofascial; post-mastectomy patients
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: A total of 61 patients who underwent total mastectomy for breast cancer with axillar lymph dissection and adjuvant radiotherapy were enrolled in this trial.
  The patients were randomized by toss of a coin to the treatment (n=30) or control (n=26) groups; of these, 48 met all study protocol requirements, including the final assessment. Inclusion criteria were: presence of functional difficulties in the shoulder area and/or upper torso on the surgical side, and 2) eligibility for physiotherapy (determined by the treating physician). Patients with recurrent disease and/or inflammatory or acute ailments were excluded. All patients gave their informed consent to participate in the study.
  The treatment group received myofascial treatment while patients in the control group received conventional therapy consisting of exercise and massage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT GROUP (Experimental): Fascial techniques were used together with the following techniques: deep massage of neck and shoulder girdle muscles; trigger point therapy; tissue scar treatment in the vicinity of the scar and directly on the scar, by stretching, breaking, pulling, as well as static and dynamic rolling; post-isometric relaxation (stretching) of shoulder and neck muscles; active release technique of the chest and shoulder; selected fascial distortion model techniques; and fascial manipulation techniques consisting of developing specific CC-center of coordination and CF-center of fusion points in the operated area and the shoulder on the same side. The exact sequence and number of procedures differed in each patient according to need as determined by prior functional examination. Before or after every of the treatment procedure treatment group patients underwent ten-minute manual lymphatic drainage in the limb on the mastectomy side.
  Interventions: Other: manual myofascial techniques
- CONTROL GROUP (Other): Treatment duration was a mean of 4 weeks. Therapy was performed daily excluding weekends and consisted of 45 minutes of individual work with an oncological physiotherapist. The control group underwent kinesiotherapeutic procedures that included various floor gymnastic exercises with gymnastic stick, balls, and/or elastic tapes, conventional massage of neck and shoulder girdle muscles and therapeutic exercises to increase ROM in the upper limb and in the chest area. Before or after every of the treatment procedure control group patients underwent ten-minute manual lymphatic drainage in the limb on the mastectomy side.
  Interventions: Other: conventional therapy consisting of exercise and massage.

INTERVENTIONS:
Other: manual myofascial techniques — Fascial techniques were used together with the following techniques: deep massage of neck and shoulder girdle muscles; trigger point therapy; tissue scar treatment in the vicinity of the scar and directly on the scar, by stretching, breaking, pulling, as well as static and dynamic rolling; post-isometric relaxation (stretching) of shoulder and neck muscles; active release technique of the chest and shoulder; selected fascial distortion model techniques; and fascial manipulation techniques consisting of developing specific CC-center of coordination and CF-center of fusion points in the operated area and the shoulder on the same side.
  Arms: TREATMENT GROUP
Other: conventional therapy consisting of exercise and massage. — Underwent kinesiotherapeutic procedures that included various floor gymnastic exercises with gymnastic stick, balls, and/or elastic tapes, conventional massage of neck and shoulder girdle muscles and therapeutic exercises to increase ROM in the upper limb and in the chest area.
  Arms: CONTROL GROUP

SUMMARY:
A total of 61 patients who underwent total mastectomy for breast cancer with axillar lymph dissection and adjuvant radiotherapy were enrolled in this trial.

The patients were randomized by toss of a coin to the treatment (n=30) or control (n=26) groups; of these, 48 met all study protocol requirements, including the final assessment. Inclusion criteria were: presence of functional difficulties in the shoulder area and/or upper torso on the surgical side, and 2) eligibility for physiotherapy (determined by the treating physician). Patients with recurrent disease and/or inflammatory or acute ailments were excluded. All patients gave their informed consent to participate in the study.

The treatment group received myofascial treatment while patients in the control group received conventional therapy consisting of exercise and massage.

DETAILED DESCRIPTION:
Treatment duration in both groups was a mean of 4 weeks. Therapy was performed daily excluding weekends and consisted of 45 minutes of individual work with an oncological physiotherapist. In the treatment group, manual myofascial techniques were used to decrease muscle tension and increase elasticity of the soft tissues in the surgical area as well as in tissues that could affect range of motion (ROM) and cause pain. Fascial techniques were used together with the following techniques: deep massage of neck and shoulder girdle muscles; trigger point therapy; tissue scar treatment in the vicinity of the scar and directly on the scar, by stretching, breaking, pulling, as well as static and dynamic rolling; post-isometric relaxation (stretching) of shoulder and neck muscles; active release technique of the chest and shoulder; selected fascial distortion model techniques; and fascial manipulation techniques consisting of developing specific CC-center of coordination and CF-center of fusion points in the operated area and the shoulder on the same side. The exact sequence and number of procedures differed in each patient according to need as determined by prior functional examination. The control group underwent kinesiotherapeutic procedures that included various floor gymnastic exercises with gymnastic stick, balls, and/or elastic tapes, conventional massage of neck and shoulder girdle muscles and therapeutic exercises to increase ROM in the upper limb and in the chest area. Both groups before or after every of the treatment procedure underwent ten-minute manual lymphatic drainage in the limb on the mastectomy side.

Patient interviews and diagnostic examinations were performed at baseline (pre-treatment) and after treatment finalization. The following variables were assessed during the diagnostic examination of the muscle length with Janda's protocol:

Pectoralis Major - pars clavicularis - the normal length of these fibers allows the patient's arm (in an extended position close to the body) to rest below the horizontal.

Pectoralis Major - pars sternocostalis - the normal length of these fibers allows the abducted the patient's arm to 90° to rest below the horizontal.

Pectoralis Major - pars abdomen - the normal length of these pectoral fibers allows the abducted the patient's arm to 150° with slight external rotation to rest in a horizontal position.

Latissimus dorsi - the normal length allows the arm to rest horizontally to the table with the lumbar spine flat on the table.

Descending part of trapezius - the length is assessed qualitatively by noting the end-feel resistance. The normal end feel is gradual rather than abrupt.

Levator scapulae - the length is assessed qualitatively by noting the end-feel resistance. The normal end feel is gradual rather than abrupt.

ELIGIBILITY:
Inclusion Criteria:

* presence of functional difficulties in the shoulder area and/or upper torso on the surgical side
* eligibility for physiotherapy (determined by the treating physician)
* signed informed consent to participate in the study.

Exclusion Criteria:

* patients with recurrent disease and/or inflammatory or acute ailments were excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
muscle length | 2 years
  muscle length with Janda's protocol
  Pectoralis Major - pars clavicularis - the normal length of these fibers allows the patient's arm (in an extended position close to the body) to rest below the horizontal.
  Pectoralis Major - pars sternocostalis - the normal length of these fibers allows the abducted the patient's arm to 90° to rest below the horizontal.
  Pectoralis Major - pars abdomen - the normal length of these pectoral fibers allows the abducted the patient's arm to 150° with slight external rotation to rest in a horizontal position.
  Latissimus dorsi - the normal length allows the arm to rest horizontally to the table with the lumbar spine flat on the table.
  Descending part of trapezius - the length is assessed qualitatively by noting the end-feel resistance. The normal end feel is gradual rather than abrupt.
  Levator scapulae - the length is assessed qualitatively by noting the end-feel resistance. The normal end feel is gradual rather than abrupt [Page et al. 2010].

SECONDARY OUTCOMES:
Active ROM in the shoulder joint on the surgical side | 2 years
  complete pathological response (pCR, pathologic Complete Response)
pathological response | 2 years
  ROM of the shoulder joint on the surgical side (flexion; extension; abduction; internal rotation; external rotation in horizontal flexion
Pain intensity | 2 years
  VAS - A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain (0) and the other end meaning the worst pain imaginable (10) . A patient marks a point ( 0 to 10) on the line that matches the amount of pain she feels."
Scar mobility | 2 years
  Made by the centimeter measure as difference of distance from the bone point, to the most limited place in the scar. It was measured in directions: cranial (distance from the ridge of the coracoid) and in the transverse direction (the distance from the xiphoidal process). The centimeter measure was the distance from the bone point (xiphoid process and coracoid), to the most limited place in the scar (which was marked on the patient's examination card so that the measurement could be repeated to the same place
Presence of the visual dysfunction of scar (retraction) and presence of the axillary web syndrome | 2 years
  Was observed presence of the visual dysfunction of scar (retraction) and presence of the axillary web syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Sławomir Marszałek, PhD, Principal Investigator — Greater Poland Cancer Centre
Locations (1):
- Greater Poland Cancer Centre, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No